CLINICAL TRIAL: NCT07274176
Title: The Effect of Graded Forced Expiration on Intraocular Pressure: A Study Using the Airofit Device
Brief Title: The Effect of Graded Forced Expiration on Intraocular Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Ali Yavuz Karahan, Professor, Uşak University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AB&AYK
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Intervention Model Description: A prospective, cross-sectional, single-visit study designed to measure the acute effect of a standardized respiratory exercise session on intraocular pressure (IOP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Forced expiration program (Experimental): The participants will be equipped with the Airofit respiratory muscle trainer and will be provided with standardised instructions on performing forced expiration manoeuvres.
  Participants will be fitted with the Airofit respiratory muscle trainer and given standardized instructions on performing forced expiration maneuvers.
  * The protocol consisted of sequentially performing forced expiration at each of the device's six predefined resistance levels (Level 1 being the lowest, Level 6 the highest).
  * The sequence for each level will be identical and as follows:
    * Exercise Phase: The participant will perform forced expiration maneuvers with the Airofit device for a duration of 5 minute at the specified resistance level.
    * Immediate Post-Exercise Measurement: Within 5 seconds of completing the exercise minute, IOP will be measured. This measurement will be labeled accordingly: T1 (after Level 1), T2 (after Level 2), up to T6 (after Level 6).
  Interventions: Other: Intraocular Pressure after forced expiration

INTERVENTIONS:
Other: Intraocular Pressure after forced expiration — The experiment will entail the acquisition of a total of seven intraocular pressure (IOP) measurements from each subject.
  * T0: Baseline (pre-intervention, resting).
  * T1: Immediately after 1 minute of forced expiration at Level 1.
  * T2: Immediately after 1 minute of forced expiration at Level 2.
  * T3: Immediately after 1 minute of forced expiration at Level 3.
  * T4: Immediately after 1 minute of forced expiration at Level 4.
  * T5: Immediately after 1 minute of forced expiration at Level 5.
  * T6: Immediately after 1 minute of forced expiration at Level 6.

SUMMARY:
The primary objective of this study is to utilize the Airofit device to systematically measure and characterize the changes in intraocular pressure across its six different levels of forced expiration. This investigation will provide crucial quantitative data on the IOP-respiratory effort relationship, enhancing our understanding of IOP dynamics during controlled respiratory stress and establishing a new, standardized paradigm for such research.

DETAILED DESCRIPTION:
Intraocular pressure (IOP) is a key physiological parameter and the primary modifiable risk factor for glaucoma. Its dynamic nature is well-documented, with fluctuations known to occur due to a variety of factors, including posture, time of day, and bodily maneuvers. The Valsalva maneuver-forced exhalation against a closed glottis-is a classic example of a physiological stressor that can cause a transient, sharp increase in IOP. This occurs due to a rise in intrathoracic and episcleral venous pressure, impeding the outflow of aqueous humor.

While the effect of a maximal Valsalva is recognized, the quantitative relationship between graded levels of expiratory force and IOP remains poorly characterized. Previous studies have been limited by the inability to precisely control and measure respiratory effort, often relying on voluntary maneuvers that lack standardization and reproducibility.

The recent advent of portable respiratory muscle trainers, such as the Airofit device, offers a novel solution to this methodological challenge. This device enables the precise application of controlled, graded resistance to expiration across multiple predefined levels.

Therefore, the primary objective of this study is to utilize the Airofit device to systematically measure and characterize the changes in intraocular pressure across its six different levels of forced expiration. This investigation will provide crucial quantitative data on the IOP-respiratory effort relationship, enhancing our understanding of IOP dynamics during controlled respiratory stress and establishing a new, standardized paradigm for such research.

Methods

Study Design: A prospective, cross-sectional, single-visit study designed to measure the acute effect of a standardized respiratory exercise session on intraocular pressure (IOP).

Participants and Recruitment

A convenience sample of 60 adult participants will be recruited from outpatient clinics of physical medicine and rehabilitation of Usak university

Participants will be provided with a full information sheet and will sign a written informed consent form prior to any study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Willing and able to provide informed consent.
* Have a best-corrected visual acuity of 6/12 or better.
* Able to understand and follow instructions for using the Airofit device.
* Have an optic nerve cup/disc ratio not exceeding 0.5, and have a c/d difference between both eyes not exceeding 0.2.
* Did not have taken any anticholinergic medication, systemic beta-blockers, or corticosteroids within the last 3 months that could affect intraocular pressure levels.

Exclusion Criteria:

* a history of intraocular surgery,
* a history of uveitis,
* a spherical refractive error exceeding 3D,
* a history of regular topical treatment other than artificial tears

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure Measurement | T0: Baseline / T1: after 1 minute of forced expiration at Level 1 /T2: after 1 minute of forced expiration at Level 2/T3: Immediately after 1 minute of forced expiration at Level 3
  The intraocular pressure will be measured in both eyes using a calibrated Tonoref III non-contact tonometry (Nidek Co., Ltd., Gamagori, Aichi, Japan) and applanation tonometry (A900 tonometer, Costruzione Strumenti Oftalmici, Firenze, Italy) by a single examiner

CONTACTS AND LOCATIONS:
Overall Officials: Ali Y Karahan, Prof., Study Chair — University of Usak
Locations (1):
- University of Usak, Uşak, Turkey (Türkiye)